CLINICAL TRIAL: NCT05671289
Title: Investigation of Urine Volatile Organic Compounds as Novel Diagnostic Biomarker in Bladder Cancer
Brief Title: Urine VOC Investigation in Bladder Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSL-004
Record Dates: First submitted 2023-01-03; First posted 2023-01-04 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-01

CONDITIONS: Bladder Cancer
Keywords: volatile organic compounds; urine; bladder cancer; GS-MS
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — 35-45 ml early morning midstream urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with confirmed bladder tumor: Patients with bladder tumor, confirmed by cystoscopy and radiology. Age ranging from 18 to 80 years old. Women of childbearing age should have negative urine pregnancy test.
  Interventions: Diagnostic Test: analysis of urine volatile organic compounds
- Healthy volunteers: Individuals with no known disease and normal urinalysis. Age ranging from 18 to 80 years old. Women of childbearing age should have negative urine pregnancy test.
  Interventions: Diagnostic Test: analysis of urine volatile organic compounds

INTERVENTIONS:
Diagnostic Test: analysis of urine volatile organic compounds — gas chromatography - mass spectrometry will be used to assess the composition of VOCs in urine samples of all participants.

SUMMARY:
The goal of this study to investigate the volatile organic compounds (VOCs) in the urine samples of both healthy individual and bladder cancer patients, using gas chromatography - mass spectrometry. Researchers aim to find a set of certain VOCs specific to bladder cancer and use this set to construct a diagnostic model that can help diagnosing bladder cancer. Participants will be asked to collect their early morning midstream urine in a predesignated container. Researchers will compare urine VOCs from bladder cancer patients and healthy individuals to see if there is any VOC whose concentration differ significantly among the two groups.

DETAILED DESCRIPTION:
Specifically, participants will be asked to collect 35-45 ml of their early morning midstream urine sample in a predesignated polytetrafluoroethylene bottle. Researcher will collect participants' health information, including their: 1)smoking history; 2)comorbidity; 3) history of past urological procedure; 4)medication; 5)pathology diagnosis after surgery, if participants have bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* bladder tumor confirmed by cystoscopy and radiology
* women of childbearing age with negative urine pregnancy test result
* willing to participate in this trial and sign the informed consent form

Exclusion Criteria:

* patient with 1) uncontrollable urinary tract infection; 2) severe systemic disease; 3) history of malignancy within the past 5 years; 4) pregnancy or lactation
* patient involved in other clinical trials
* other situations researcher considered to be ineligible for this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatients with confirmed bladder tumor, present in first affiliated hospital of Xi'an jiaotong university during the recruitment phase, are recruited. Healthy volunteers are recruited outside the hospital with invitations to participate.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Urine volatile organic compounds composition of all urine samples | immediately after GC-MS analysis has been finished
  Data derived from mass spectrums of GC-MS measurement of VOC components in urine samples, including VOC components identified comparing obtained data to those in public GC-MS database and the absolute concentration of VOCs identified.

SECONDARY OUTCOMES:
Pathological diagnosis of bladder tumor patients enrolled | Immediately after the release of pathological examination reports by pathology department in the First affiliated hospital of Xi'an jiaotong university
  Staging of bladder cancer using American Joint Committee on Cancer (AJCC) TNM system and histology of tumor tissue will be collected, if patient has received surgery during hospitalization. Concerning bladder tumor patients only.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Fan, MD, Study Director — First affiliated hospital of Xian jiaotong university
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided